CLINICAL TRIAL: NCT04659070
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Phase 3 Trial to Evaluate the Efficacy and Safety of Co-administrated Ezetimibe/Rosuvastatin and Telmisartan in Patients With Essential Hypertension and Primary Hypercholesterolemia
Brief Title: To Evaluate the Efficacy and Safety of Co-administrated Ezetimibe/Rosuvastatin and Telmisartan in Patients With Essential Hypertension and Primary Hypercholesterolemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL-CDP-301
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Primary Hypercholesterolemia; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Rosuvastatin Calcium; Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental : Ezetimibe / Rosuvastatin + Telmisartan (Experimental): Ezetimibe 10mg / Rosuvastatin 20mg + Telmisartan 80mg PO, Once daily for 8 weeks
  Interventions: Drug: Experimental : Ezetimibe / Rosuvastatin + Telmisartan
- Active comparator1 : Ezetimibe / Rosuvastatin (Active Comparator): Ezetimibe 10mg / Rosuvastatin 20mg PO, Once daily for 8 weeks
  Interventions: Drug: Active comparator1 : Ezetimibe / Rosuvastatin
- Active comparator2 : Telmisartan (Active Comparator): Telmisartan 80mg PO, Once daily for 8 weeks
  Interventions: Drug: Active comparator2 : Telmisartan

INTERVENTIONS:
Drug: Experimental : Ezetimibe / Rosuvastatin + Telmisartan — Ezetimibe 10mg / Rosuvastatin 20mg + Telmisartan 80mg PO, Once daily for 8 weeks
  Arms: Experimental : Ezetimibe / Rosuvastatin + Telmisartan
Drug: Active comparator1 : Ezetimibe / Rosuvastatin — Ezetimibe 10mg / Rosuvastatin 20mg PO, Once daily for 8 weeks
  Arms: Active comparator1 : Ezetimibe / Rosuvastatin
Drug: Active comparator2 : Telmisartan — Telmisartan 80mg PO, Once daily for 8 weeks
  Arms: Active comparator2 : Telmisartan

SUMMARY:
This study is a multicenter, Randomized, double-blind, acitve-controlled, Phase 3 Clinical Trial in 8 weeks for screening, twice Investigational product administer, Follow up visit.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of Co-administrated Ezetimibe/Rosuvastatin and Telmisartan in patients with essential hypertension and primary hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female aged 19 to 79 years of age
2. a patient with congenital hypertension and hypercholesterolemia capable of administering medicines for Clinical trials planned for this clinical trial, with the discontinuation of existing therapeutic drugs according to the section.
3. A person who meets the following criteria at the time of screening (visit 1)

   * MSSBP < 180mmHg and MSDBP < 110mmHg
   * LDL-C ≤ 250 mg/dL and TG < 400 mg/dL (based on organ clinical laboratory testing)
4. A person who agrees to contraception through a medically permitted contraception method during a clinical trial period.

   * Possible pregnant female test subjects: intrauterine device (IUD) or IUS (Intrauterine system), intractorine defections, double-blocking method (complex use of blocking methods such as male condoms, female condoms, uterine cervical caps, contraceptive diaphragm, contraceptive sponges)
   * Male test subjects with potential pregnant spouses (including partners): hormonal contraception, intrauterine device (IUD) or IUS (Intrauterine system), intraperitoneal failure, double-blocking (male condom, female condom, uterine cervical cap, contraceptive diaphragm, and contraceptive blocking)
5. Patients who have agreed in writing to voluntarily participate in this clinical trial

Randomized(Visit 2) criteria

1. If the blood pressure measured at the time of random assignment is as follows:

   - 140mmHg ≤ MSSBP < 180mmHg and MSDBP < 110mmHg However, patients with diabetes or chronic neuropathy: 130mmHg ≤ MSSBP < 180mmHg (In the case of chronic neuropathy patients, albuinuria or proteinuria history is confirmed until the time of random assignment.)
2. Therapeutic Lifestyle Change (TLC) after Visit 1 A person whose LDL-C and TG values correspond to the following group-specific criteria (NCEP ATP III guideline) as the basis for organ testing at the time of random assignment.

   * Group1 cardiovascular risk factor : 0~1, LDL-C(mg/dL) : 160-250, TG(mg/dL) : < 400
   * Group2 cardiovascular risk factor : 2 ≤, 10 year risk : < 10% LDL-C(mg/dL) : 160-250 TG(mg/dL) : < 400 cardiovascular risk factor : 2 ≤, 10% ≤ 10 year risk ≤ 20%, LDL-C(mg/dL) : 130-250 TG(mg/dL) : < 400
   * Group3 coronary artery disease or equivalent (20% < 10 year risk), LDL-C(mg/dL) : 100-250 TG(mg/dL) : < 400
3. A person who does not have any inappropriate items when re-checking the selection/excluding criteria at the time of random assignment.

(except items that apply only to screening)

Exclusion Criteria:

1. A person suspected of secondary hypertension or secondary hypertension (aortic stenosis, hyperaldosterone haemorrhage, renal vein stenosis, sacrosanctal hypertension, chrome-friendly cell species, Cushing syndrome, polycystic neuropathy, etc.)
2. Secondary dyslipidemia patients (neurological syndrome, dysplasia, closed liver disease, Cushing syndrome, etc.)
3. Standing low blood pressure patient with symptoms
4. Clinically meaningful ventricular tachycardia, atrial fibrillation, atrial fibrillation, or other arrhythmia patients that the tester has determined to be clinically meaningful.
5. Persons with non-post-closing myocardial disease, severe closed coronary artery disease, aortic stenosis, hemodynamically meaningful aortic valve or mitral valve stenosis.
6. Patients with severe heart failure (NYHA class III: Symptoms due to mild exercise/classIV: Symptoms even when stabilized)
7. A person who has one or more of the following forces within the last six months based on a screening visit (visit 1):

   * Those who have received ischemic heart disease (unstable angina, myocardial infarction), peripheral vascular disease, percutaneous coronary artery extension or coronary artery bypass treatment, etc.
   * Patients with severe cerebrovascular disorders (brain stroke, cerebral infarction, cerebral hemorrhage, routine ischemia, etc.)
8. A person with a history of gastrointestinal diseases (such as Crohn's disease, ulcers, etc.) and surgery (except simple appendectomy or hernia surgery) that can affect the absorption, distribution, metabolism, and excretion of drugs.
9. Patients with gastrointestinal diseases such as active gastritis or duodenal ulcer within one year of screening
10. A person who has a history of muscle toxicity to fibromyalgia, myopathy, rhabdomyolysis, history of hereditary muscle disease or family history, and past HMGCoA reducing enzyme inhibitor or fibrate-related drugs.
11. Patients with parathyroidism
12. Patients with shock
13. Patients with biliary obstruction or bile congestion
14. Patients with hereditary vascular edema
15. Patients with a history of vascular edema during ACE inhibitor or Angiotensin II receptor antagonist treatment.
16. Patients with chronic inflammatory diseases who need continuous anti-inflammatory treatment
17. Patients with autoimmune diseases, connective tissue diseases
18. Those who have a history of moderate degree or malignant retinopathy (i.e., retinal bleeding, vision impairment, retinal micro aneurysm) within the previous six months based on a screening visit (visit 1)
19. On the basis of a screening visit (visit 1) a person with malignancy, including leukemia and lymphoma, was evaluated as Complete Response (but not recurrent within at least two years from the screening date, or a malignant tumor that occurred within the minimum two years of the screening, is the only basal cell carcinoma or squamous skin cell carcinoma (Square).
20. Patients who have run out of blood or sodium due to high doses of diuretics, dietary salinity, diarrhea and vomiting.
21. The following institutional clinical laboratory test results (screening criteria) are available:

    * Patients with active liver disease and severe liver disorder (unknown continuous serum AST, elevated or serum ALT, person with AST more than three times the normal upper limit)
    * a person whose CPK (creatine phosphokinase) level is more than twice the normal upper limit.
    * Creatine clearance (CLcr) < 30mL/min or eGFR < 30ml/min/1.73m2.
    * a person with low potassium haemorrhage (less than 3.5 mmol/L) or high potassium haemorrhage (greater than 5.5 mmol/L)
    * Unregulated diabetics (HbA1c > 9.0%)
    * Unregulated thyroid dysfunction with a TSH level of 1.5 times or more than the normal upper limit
22. In case of the following allergic and hypersensitive history:

    * someone with drug allergy-response anaphylaxis or hepatotoxicity.
    * Angiotensin II receptor blocker family drug or HMG-CoA reducing enzyme inhibitor
    * A person who has overreacted to a clinical trial drug or is hypersensitive to the composition of a clinical trial drug
    * A person who has genetic problems such as galactose intolerance, Lap lactase deficiencies, or glucose-galactose malabsorbtion.
23. A person who is administering a prohibited drug in this clinical trial or is expected to be administered during the clinical trial period.
24. Those who showed a difference of SBP ≥ 20 mmHg and DBP ≥10 mmHg in three consecutive measurements at least two minutes apart on each arm during a screening visit (visit 1)
25. Patients who cannot stop anti-hypertensive drugs or lipid-control drugs that were being administered during a screening visit (visit 1) during the clinical trial period.
26. Those who have or are suspected of drug or alcohol abuse within one year prior to the screening visit (visit 1)
27. Pregnant or breastfeeding women
28. A person who has received another clinical trial medication within three months of the first administration of the clinical trial medication in this clinical trial (if he/she has not administered the clinical trial medication or has participated in non-release observation research, he/she may register).
29. A person who is deemed unfit by the tester (the physician in charge) to participate in this clinical trial

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-05-19 (Estimated); Study Completion 2022-05-19 (Estimated)

PRIMARY OUTCOMES:
Mean sitting systolic blood pressure (MSSBP) | baseline, week 8
  MSSBP change at week 8 compared to baseline, experimental, active comparator1
Low density lipoprotein cholesterol (LDL-C) | baseline, week 8
  LDL-C change at week 8 compare to baseline, experimental, active comparator2

SECONDARY OUTCOMES:
Mean sitting systolic blood pressure (MSSBP) | baseline, week 4
  MSSBP change at week 4 compare to basline, experimental, active comparator1
Mean sitting diastolic blood pressure (MSDBP) | baseline, week 4, week 8
  MSDBP change at week 4, 8 compare to baseline, experimental, active comparator1
the rate of patients who have reached their target blood pressure | week4, week8
  The rate of patients who have reached their target blood pressure in experimental and active comparator1 at 4 or 8 weeks after administration of clinical trial medications (Average left blood pressure < 140/90mmHg, diabetic or chronic renal disease (only for patients with chronic renal disease with albu manure or proteinuria history) Average left and right blood pressure / 130/80mmHg)
Percentage of LDL-C change | baseline, week4
  Percentage of LDL-C change at week 4 compare to baseline, experimental, active comparator2
LDL-C change | baseline, week4, week8
  LDL-C change at week 4, 8 compare to baseline, experimental, active comparator2
Achievement rate of LDL-C treatment goals | week4, week8
  Achievement rate of LDL-C treatment goals in accordance with NCEP ATP III criteria at 4 and 8 weeks after administration of clinical trial medications, experimental, active comparator2 (Group1 : < 160mg/dL, Group 2: < 130mg/dL, Group 3: < 100mg/dL)
Percentage of lipid indicators change | baseline, week4. week8
  Percentage of lipid indicators(TC, HDL-C, TG, LDL-C/HDL-C, TC/HDL-C, non-HDL-C, Apo B) change at week 4, 8 compare to baseline, experimental, active comparator2
Lipid indicators chage | basline, week4, week8
  Lipid indicators(TC, HDL-C, TG, LDL-C/HDL-C, TC/HDL-C, non-HDL-C, Apo B) change at week 4, 8 compare to baseline, experimental, active comparator2

CONTACTS AND LOCATIONS:
Locations (1):
- Daegu Catholic Univ Medical Center, Daegu, South Korea